CLINICAL TRIAL: NCT04344860
Title: Prospective, Randomized Trial Comparing Recombinant Von Willebrand Factor (rVWF) Plus Tranexamic Acid vs. rVWF Alone to Reduce Postpartum Hemorrhage in Women With Von Willebrand Disease: The VWD-WOMAN Trial
Brief Title: Prevent Postpartum Hemorrhage in Women With Von Willebrand Disease: The VWD-WOMAN Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nicoletta C Machin (Other)
Responsible Party: Sponsor-Investigator, Nicoletta C Machin, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY20030186
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Von Willebrand Diseases; Postpartum Hemorrhage
MeSH Terms: conditions — von Willebrand Diseases; Postpartum Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Randomized, Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- rVWF plus TA (Active Comparator): Subjects randomized to this arm will receive recombinant von Willebrand factor 80 IU/kg IV within 5-10 minutes of delivery (or epidural anesthesia) plus Tranexamic Acid 1 gm IV within 3 hours of delivery; and recombinant Von Willebrand factor 80 IU/kg on day 1 and day 2 postpartum.
  Interventions: Drug: Recombinant Von Willebrand factor; Drug: Tranexamic Acid Injection [Cyklokapron]
- rVWF alone (Active Comparator): Subjects randomized to this arm will receive recombinant von Willebrand factor 80 IU/kg IV within 5-10 minutes of delivery (or epidural anesthesia); and recombinant Von Willebrand factor 80 IU/kg on day 1 and day 2 postpartum.
  Interventions: Drug: Recombinant Von Willebrand factor

INTERVENTIONS:
Drug: Recombinant Von Willebrand factor — Recombinant Von Willebrand factor(Vonvendi) is an intravenous therapy that replaces missing VWF to restore hemostasis and reduce bleeding with surgery or delivery.
  Other Names: rVWF, Vonvendi
Drug: Tranexamic Acid Injection [Cyklokapron] — Tranexamic acid (Cyclokapron) is an intravenous anti-fibrinolytic therapy that prevents clot breakdown and reduces bleeding with surgery or delivery.
  Other Names: TA, Cyclokapron
  Arms: rVWF plus TA

SUMMARY:
This is a single-center randomized phase III clinical trial, the VWD-Woman Trial, in which 20 pregnant subjects with von Willebrand disease (VWD), defined as VWF ristocetin co-factor activity (VWF:RCo) <0.50 IU/ml (historic) and previous history of bleeding are enrolled. Subjects will include women with VWD age 18 years and older, excluding those who have a bleeding disorder other than VWD. Once enrolled, subjects who meet all of the inclusion and none of the exclusion criteria will be randomized to recombinant Von Willebrand factor (rVWF, Vonvendi ®) with Tranexamic Acid (TA, Cyclokapron®); or recombinant Von Willebrand factor (rVWF, Vonvendi®) alone to prevent postpartum hemorrhage after vaginal or caesarean delivery. The primary endpoint is quantitative blood loss (QBL) by a labor suite nurse at delivery. Secondary endpoints include safety assessment for postpartum lochial blood loss by Pictorial Blood Assessment Chart (PBAC), transfusion, blood products, thromboembolic events, and hysterectomy within 21 days; and mechanism of PPH reduction by VWF assays (VWF:RCo, VWF:Ag, VIII:C), fibrinogen, and d-dimer. Blood draws are at 5 time points, including at 36 weeks' gestation (screening), on admission for childbirth, and at 1 day, 2 days, and 21 days after delivery. The VWD-Woman Trial is considered greater than minimal risk as study drugs are given at delivery and special coagulation studies are obtained.

DETAILED DESCRIPTION:
The purpose of this 8-week single center, randomized, open-label phase III trial to compare recombinant von Willebrand factor (rVWF, Vonvendi®)) plus tranexamic acid (TA, Cyclokapron®) vs. rVWF alone to prevent postpartum hemorrhage (PPH) in women with Von Willebrand disease (VWD). VWD is an inherited bleeding disorder that occurs in 1% of the population. It is caused by deficient or defective von Willebrand factor (VWF). Treatment at delivery is with VWF concentrate, based on U.S. and European guidelines, and as DDAVP, a non-VWF protein, is contraindicated as it may cause hyponatremia (low salt) and seizures due to fluid replacement at delivery. Yet, blood loss is 1.5-fold greater in VWD than non-VWD controls. The investigators believe this is due to physiologic (protective) fibrinolysis (clot breakdown) in the first 3 hours after delivery, which may protect controls from excess clotting after delivery, but which may increase bleeding in subjects with VWD. PPH a significant cause of maternal morbidity and mortality in women. PPH is defined as >1000 ml within the first 24 hours of vaginal or cesarean delivery. PPH peaks in the first 2-3 hours postpartum, a time during which there is early activation of the fibrinolytic system, with a 2-fold increase TPA (tissue plasminogen activator). So while uterine atony is the major cause of PPH, accounting for 63% of PPH cases, but in 37% of cases, uterotonic agents fail.

TA is an anti-fibrinolytic therapy (prevents clot breakdown) which reduces bleeding and prevents clot breakdown in surgery, trauma, and in controls at delivery, if it is given within 3 hours of delivery. In the WOMAN trial, a large trial of over 10,000 women without bleeding disorders, TA was safe and effective in reducing PPH when given intravenously (in a vein) within 3 hours of vaginal or cesarean delivery. As TA is approved by the US. Food and Drug Administration (FDA) to treat and prevent bleeding in VWD, the investigators propose to study rVWF plus TA vs. VWF alone to reduce PPH in subjects with VWD. This is a pilot study to determine if recruitment, randomization, and study drug administration can be performed successfully, and shows preliminary safety and efficacy in subjects with VWD. rVWF (Vonvendi®) will be administered by intravenous infusion before delivery and on day 1 and day 2 postpartum. Tranexamic acid (Cyclokapron®) will be administered by intravenous infusion within 3 hours postpartum. Randomization will be at delivery to either rVWF at delivery and on day 1 and day 2 postpartum, plus TA within three hours postpartum; or rVWF alone at delivery and on day 1 and day 2 postpartum.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant females >= 18 years of age
2. Confirmed VWD, as defined by VWF:RCo < 0.50 IU/dL and previous history of bleeding
3. Willingness to have blood drawn
4. Willing to be randomized to one of two treatments at delivery and for 2 days postpartum.
5. Willing to keep a diary for 3 weeks of postpartum bleeding by pictorial assessment chart (PBAC) and any blood products, transfusion, or medications taken.
6. Willing to return at 21 days for final blood draw and review of diary.

Exclusion Criteria:

1. Any bleeding disorder other than VWD; or past thrombotic disease of other bleeding disorders.
2. Previous thrombosis, cardiac disease, congestive failure, arrhythmia, hypertension, MI, or stroke.
3. Platelet count < 100,000/ ul.
4. Past allergic reaction to VWF or tranexamic acid.
5. Surgery within the past 8 weeks.
6. Inability to comply with study protocol requirements.
7. Concomitant use of antiplatelet drugs, anticoagulants, or NSAIDs. Aspirin will be allowed for preeclampsia prevention.
8. Treatment with DDAVP, cryoprecipitate, whole blood, plasma or plasma derivatives containing substantial quantities of VWF within 5 days of study.
9. History of renal disease.
10. Inability to comply with study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicoletta Machin, DO, Principal Investigator — University of Pittsburgh
Locations (1):
- Hemophilia Center of Western PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The IPD to be shared include individual bleeding data (EBL, PBAC); hemostasis agents (blood product usage, transfusion, other medications); and VWF assays (VWF:RCo, VWF:Ag, FVIII:C) and coagulation assays (fibrinogen, d-dimer).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 12 months of trial completion.
Access Criteria: Qualified investigators will have access to data and biospecimens, consistent with data sharing policies and applicable laws, and upon receipt of a Research Materials Distribution Agreement, data will be transferred by secure transfer through the GSPH portal website.

REFERENCES:
- [Background] Ragni MV, Machin N, James AH, Seaman CD, Malec LM, Kessler CM, Konkle BA, Kouides PA, Neff AT, Philipp CS, Brooks MM. Feasibility of the Von Willebrand disease PREVENT trial. Thromb Res. 2017 Aug;156:8-13. doi: 10.1016/j.thromres.2017.05.022. Epub 2017 May 25. PMID 28577390
- [Background] Ragni MV. Blood volume-based von Willebrand factor to prevent postpartum hemorrhage in von Willebrand disease. Blood Adv. 2017 Apr 25;1(11):703-706. doi: 10.1182/bloodadvances.2017005090. eCollection 2017 Apr 25. PMID 29296713
- [Background] Ragni MV. Case-based discussion on the implications of exogenous estrogens in hemostasis and thrombosis: the hematologist's view. Hematology Am Soc Hematol Educ Program. 2019 Dec 6;2019(1):152-157. doi: 10.1182/hematology.2019000022. PMID 31808846
- [Derived] Machin NC, Brooks MM, Vehec D, Ivanco D, Lawryk B, Seaman CD, Xavier F, Shiva S, Verdoni A, Ragni MV. Impact of tranexamic acid on postpartum hemorrhage in type 1 von Willebrand disease treated with recombinant VWF. Blood Adv. 2025 Dec 9;9(23):6031-6039. doi: 10.1182/bloodadvances.2025017046. PMID 40902088

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened and enrolled during routine clinic visits at the Hemophilia Center of Western Pennsylvania, with delivery planned at UPMC Magee-Womens Hospital in Pittsburgh, Pennsylvania. The study was approved by the University of Pittsburgh Biomedical Institutional Review Board April 28, 2021, and between June 4, 2021 and May 17, 2024, 20 patients were enrolled.
Period: Overall Study
Arm/Group | rVWF plus TA | rVWF alone
Started | 10 | 10
Completed (103 screened → 40 eligible → 20 randomized (10 each group). Reasons for non-enrollment: delivery outside site, diagnosis not verified, declined participation.) | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rVWF plus TA | rVWF alone | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (5.2) | 28.8 (5.3) | 29.0 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Ferritin [Mean (Standard Deviation); unit: ng/mL] — Abnormally low ferritin is defined as <50 μg/L in the context of pregnancy.
  ng/mL | 18 (11.1) | 13.5 (6.5) | 15.8 (9.1)
Third Trimester Hemoglobin [Median (Standard Deviation); unit: dL] — Hemoglobin at the third-trimester screening visit.
  dL | 12.1 (0.9) | 11.8 (1.0) | 11.9 (0.9)
VWF:Ag 3rd trimester [Median (Standard Deviation); unit: IU/mL] | 1.9 (1.1) | 1.4 (1.1) | 1.7 (1.1)
Number of participant with type 1 von Willebrand disease [Count of Participants; unit: Participants] — von Willebrand subtype based on historic characterization (type 1, type 2, type 3). Type 1 von Willebrand disease (VWD) was confirmed per diagnostic criteria based on reduced plasma VWF antigen and/or VWF activity levels (typically <50 IU/dL) with concordant bleeding phenotype and family history, consistent with 2021 ISTH classification guidelines.
  Participants | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Volume of Quantitative Blood Loss at Delivery
Description: Blood loss at delivery by standard QBL measured for 6 hours postpartum by the labor and delivery nursing staff.
Time Frame: 6hrs
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | rVWF plus TA | rVWF alone
Number analyzed (Participants) | 10 | 10
mL | 727.0 (802.5) | 539.7 (355.08)

2. Secondary Outcome: Blood Loss Postpartum by Pictorial Bleeding Assessment Chart (PBAC)
Description: Blood loss postpartum by pictorial bleeding assessment chart (PBAC).
  Participants record the degree of saturation of sanitary products and the presence of clots.
  Total PBAC scores range from 0 to >500, with higher scores indicating heavier menstrual bleeding.
  A score ≥100 is conventionally consistent with heavy bleeding.
  Each sanitary product is assigned a score reflecting the amount of blood loss:
  Pads: 1 (point) for lightly stained, 5 for moderately soiled, 20 for fully soaked Tampons: 1 for lightly stained, 5 for moderately soiled, 10 for fully soaked Clots: 1 point for small (<1 cm), 5 for large (>1 cm) Daily scores are summed to produce a total cycle PBAC score. Subscale items (pads and clots) were summed to obtain a total PBAC score.
Time Frame: 21 days
Population: One subject in the rVWF+ TA arm did not complete a PBAC diary and was excluded from this exploratory analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | rVWF plus TA | rVWF alone
Number analyzed (Participants) | 9 | 10
Scores on a scale | 467.1 (442.0) | 344.8 (315.5)

3. Secondary Outcome: Number of Blood Products Used
Description: Number of transfused blood products determined by electronic medical record review and patient diary.
Time Frame: 21 days
Population: All subjects were included in this analysis.
Measure: Number; unit: Number of transfused blood products
Arm/Group | rVWF plus TA | rVWF alone
Number analyzed (Participants) | 10 | 10
Number of transfused blood products | 0 | 0

4. Secondary Outcome: Concentration of Von Willebrand Factor
Description: Plasma levels of von Willebrand Factor antigen (VWF:Ag) and activity (VWF:RCo) measured during the peripartum period. Higher concentrations indicate greater clotting factor activity.
Time Frame: 21 days
Population: All randomized participants (N=20; 10 per arm) were included in the analysis. For von Willebrand factor laboratory outcomes (VWF:Ag, VWF:RCo), not all participants contributed data at every time point due to missed blood draws. Specifically, one participant in the rVWF+TXA arm had missing values at 48 hours postpartum and at 21 days postpartum. Therefore, the analysis population for those time points is n=9 in the rVWF+TXA arm and n=10 in the rVWF-alone arm.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | rVWF plus TA | rVWF alone
Number analyzed (Participants) | 10 | 10
IU/mL
  Third trimester VWF:Ag | 1.89 (1.1) | 1.41 (0.6)
  Admission VWF:Ag | 2.20 (1.1) | 2.00 (1.0)
  24h postpartum VWF:Ag | 3.3 (0.9) | 3.4 (1.3)
  48h postpartum VWF:Ag: number analyzed (Participants) | 9 | 10
  48h postpartum VWF:Ag | 4.0 (1.2) | 3.5 (0.9)
  21 days postpartum VWF:Ag: number analyzed (Participants) | 9 | 10
  21 days postpartum VWF:Ag | 0.9 (0.7) | 0.9 (0.3)
  Third trimester VWF:RCo | 1.00 (0.5) | 1.08 (0.7)
  Admission VWF:RCo | 0.97 (0.5) | 1.1 (0.6)
  24h postpartum VWF:RCo | 1.9 (0.9) | 2.2 (0.9)
  48h postpartum VWF:Rco | 2.3 (0.6) | 2.1 (0.8)
  21 days postpartum VWF:RCo | 0.5 (0.2) | 0.5 (0.2)

ADVERSE EVENTS:
Time Frame: From enrollment until the end of follow up at 21 days
Arm/Group | rVWF plus TA | rVWF alone
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
There are several limitations of this study. First, the small sample size and pilot nature of this study restrict the generalizability of the findings. Further, as findings in type 1 VWD may not predict those with more severe disease, future studies should include pregnant females with type 2 and 3 VWD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/60/NCT04344860/Prot_SAP_000.pdf